CLINICAL TRIAL: NCT04473170
Title: Adaptive Open-label Study Evaluating the Safety and Efficacy of Autologous Non- Hematopoietic Peripheral Blood Stem Cells Therapy in COVID-19 Outbreak in Abu Dhabi, 2020 (SENTAD-COVID Study)
Brief Title: Study Evaluating the Safety and Efficacy of Autologous Non-Hematopoietic Peripheral Blood Stem Cells in COVID-19
Acronym: SENTAD-COVID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abu Dhabi Stem Cells Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT.001.1.0.SENTAD-COVID
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: COVID-19; Non-Hematopoietic Peripheral Blood Stem Cells
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Parallel assignment involving two groups of participants:
  * Group A (Experimental arm): Autologous Non-Hematopoietic Peripheral Blood Stem Cells (NHPBSC) therapy as add-on COVID-19 standard care.
  * Group B (No investigational intervention arm): COVID-19 standard care.
Masking Description: None (open-label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Autologous Non-Hematopoietic Peripheral Blood Stem Cells (NHPBSC) therapy as add-on COVID-19 standard care.
  Interventions: Biological: Autologous Non-Hematopoietic Peripheral Blood Stem Cells (NHPBSC)
- Group B (Active Comparator): COVID-19 Standard care.
  Interventions: Drug: COVID-19 standard care

INTERVENTIONS:
Biological: Autologous Non-Hematopoietic Peripheral Blood Stem Cells (NHPBSC) — SENTAD-COVID Study intervention consists of Autologous Non-Hematopoietic Peripheral Blood Stem Cells (NHPBSC) therapy through jet nebulization in addition to standard care. The NHPBSC were characterized as CD90+, CD133+, Oct-4+ (pluripotent markers), and CD45-, CD71-, based on multiparameter flow cytometry.
  Other Names: UAECell19
  Arms: Group A
Drug: COVID-19 standard care — UAE National Guidelines for Clinical Management and Treatment of COVID-19.
  Other Names: Current COVID-19 standard care in the UAE
  Arms: Group B

SUMMARY:
SENTAD-COVID Study is an adaptive, prospective, multicentric, open-label, and randomized controlled clinical trial involving hospitalized adult patients with confirmed coronavirus disease 2019 (COVID-19) infection during the outbreak in Abu Dhabi, 2020. The patients were randomly allocated in a parallel assignment involving two groups of participants: Group A (Experimental arm): autologous non-hematopoietic peripheral blood stem cells (NHPBSC) therapy as add-on COVID-19 standard care, or Group B (No investigational intervention arm): COVID-19 standard care. Standard care is defined as per the "UAE National Guidelines for Clinical Management and Treatment of COVID-19". SENTAD-COVID Study was conducted in the Sheikh Khalifa Medical City (SKMC) of Abu Dhabi, as Primary Care Clinical Trial Unit, while the cell processing and investigational product formulation were completed by Abu Dhabi Stem Cells Center (ADSCC), according to Good Laboratory Practices (GLPs) and Good Manufacturing Practices (GMPs).

DETAILED DESCRIPTION:
Group A patients received autologous NHPBSC therapy through jet nebulization, in addition to the standard care, while Group B (No investigational intervention arm) received only the UAE approved standard care. The primary endpoints were the safety and efficacy assessment, measured as Adverse Reactions (ARs) incidence [according to World Health Organization - Uppsala Monitoring Centre (WHO-UMC) causality assessment system], rate of mortality within 28-days, and the time to clinical improvement of 2 points on a seven-category ordinal scale or discharge from the Hospital, whichever came first. Immune response profile, acute-phase serum markers, and coagulation testing profile were evaluated as well, before treatment (baseline - Day 0), at Day 14, and Day 21 (in patients with early response, defined as 2 points of difference in the clinical critical treatment index within 7 days of treatment, the assessment will be performed at Day 7). The trial was approved by the institutional ADSCC Research Ethics Committees (REC), and the Emirates Institutional Review Board (IRB) for COVID-19 Research and the written informed consent was obtained from all patients or from the patient's legal representative if the patient was too unwell to provide consent. SENTAD-COVID Study was conducted in accordance with the principles of the Declaration of Helsinki and the Good Clinical Practice (GCP) Guidelines of the International Conference on Harmonization (ICH). The authors were responsible for designing the trial and for compiling and analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* RT-PCR Laboratory confirmation of COVID-19.
* Male or female aged ≥ 18 years.
* Interstitial lung change ≥ 3 judged by "Lungs Lobar based scoring" according to computed tomography (CT) scans.
* Hospitalized and symptomatic patients, referring one or more of the following symptoms (fever, cough, or shortness of breath), in association with (at least one): tiredness, runny nose, headache, sore throat, chills, muscle pain, or new loss of taste or smell).
* Ability to comply with test requirements and peripheral blood stem cells collection.
* The patient or legal representative agrees to participate in the study, and signs the SENTAD-COVID Study informed consent form.

Exclusion Criteria:

* Pediatric patients (aged < 18 years).
* Diagnosis of any kind of shock.
* Organ transplants in the past 3 months.
* Patients receiving immunosuppressive therapy.
* Diagnostic of Hepatitis B Virus (HBV) infection.
* Diagnostic of Human Immunodeficiency Virus (HIV) infection or Acquired Immunodeficiency Syndrome (AIDS).
* Current diagnosis of cancer.
* History of malignancies in the past 5 years.
* Pregnant or lactating women.
* Have participated in other clinical trials in the past 3 months.
* Inability to comply with test requirements and peripheral blood stem cells collection.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Adverse reactions incidence. | Day 0 - 28
  Proportion of participants with treatment-related Adverse Event as assessed by CTCAE v5.0.
Rate of mortality within 28-days. | Day 0 - 28
  Incidence of deaths within 28-days in enrolled patients.
Time to clinical improvement on a seven-category ordinal scale. | Day 0 - 28
  Days from administration of the Investigational Product to improvement of seven-category ordinal scale by at least 2 points.

SECONDARY OUTCOMES:
Assessment of the immune response profile. | Days 0, 14, and 28
  Immune response profile characterized according the biomarkers: CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD20, CD25, CD27, CD28, CD38, CD45, CD45RA, CD45RO, CD56, CD57, CD66b, CD123, CD127, CD161, CD294, CCR4, CCR6, CCR7, CXCR3, CXCR5, HLA-DR, IgD, and TCRγδ, for the identification of immune cells and subsets analysis; and the humoral Immune profile: IgG, IgA, IgM levels.
Assessment of acute-phase serum markers. | Days 0, 14, and 28
  Complete Blood Counts (CBC), Acute phase proteins and Inflammatory markers: CRP, ESR, LDH, Procalcitonin (PCT), Ceruloplasmin, Haptoglobin, alpha 1 antitrypsin, IL-6, ferritin C3, PT, fibrinogen and D-dimer.

CONTACTS AND LOCATIONS:
Overall Officials: Yendry Ventura Carmenate, M.D., Principal Investigator — Abu Dhabi Stem Cells Center (ADSCC)
Locations (1):
- Abu Dhabi Stem Cells Center, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castillo Aleman YM, Villegas Valverde CA, Ventura Carmenate Y, Abdel Hadi L, Rivero Jimenez RA, Rezgui R, Alagha SH, Shamat S, Bencomo Hernandez AA. Viability assessment of human peripheral blood-derived stem cells after three methods of nebulization. Am J Stem Cells. 2021 Oct 15;10(4):68-78. eCollection 2021. PMID 34849303
- [Derived] Ventura-Carmenate Y, Alkaabi FM, Castillo-Aleman YM, Villegas-Valverde CA, Ahmed YM, Sanna P, Almarzooqi AA, Abdelrazik A, Torres-Zambrano GM, Wade-Mateo M, Quesada-Saliba D, Abdel Hadi L, Bencomo-Hernandez AA, Rivero-Jimenez RA. Safety and efficacy of autologous non-hematopoietic enriched stem cell nebulization in COVID-19 patients: a randomized clinical trial, Abu Dhabi 2020. Transl Med Commun. 2021;6(1):25. doi: 10.1186/s41231-021-00101-5. Epub 2021 Nov 3. PMID 34746417